CLINICAL TRIAL: NCT00001982
Title: Natural History of Chronic Hepatitis C Among Volunteer Blood Donors
Brief Title: History of Hepatitis C in Volunteer Blood Donors
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930159; 93-DK-0159
Record Dates: First submitted 2000-01-21; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Hepatitis C
Keywords: Aminotransferases; Anti-HCV; Blood Donors; HCV RNA; Hepatitis C; Liver Biopsy; Serum Aminotransferases; Transfusion
MeSH Terms: conditions — Hepatitis C

SUMMARY:
Hepatitis C is a disease of the liver caused by the Hepatitis C Virus (HCV). Patients with hepatitis C may feel well and show no signs or symptoms of being ill. However, researchers would like to study the long-term effects of this disease.

Volunteer blood donors diagnosed with chronic hepatitis C viral (HCV) and various levels of liver enzyme activity will be offered a complete medical evaluation and liver biopsy. The tests will enable researchers to provide the patients with an idea of how severe their liver disease is. The virus and patient will be studied in order to understand why patients with hepatitis C develop different levels of liver damage.

DETAILED DESCRIPTION:
A selected sample of volunteer blood donors with chronic hepatitis C viral (HCV) infection and various levels of serum aminotransferase activity will be offered a complete medical evaluation and liver biopsy to determine the severity of their liver disease. Various virological and host factors will be studied in an attempt to determine why patients with HCV infection develop differing degrees of liver disease.

ELIGIBILITY:
Patients with chronic hepatitis C.

Age 18 to 70 years, male or female.

HCV infection indicated by the presence of anti-HCV (by ELISA and recombinant immunoblot assay [RIBA]).

Written informed consent.

Women must not be pregnant.

Patients must not have significant systemic illnesses other than liver disease, including congestive heart failure, renal failure, uncontrolled diabetes mellitus.

Patients must not have antiviral or immunosuppressive therapy within the last 6 months.

Patients must not have HIV infection.

Patients must not have contraindications to liver biopsy (mainly clotting abnormality (coumadin therapy, platelet count less than 50,000/cubic millimeter, prothrombin time more than 4 seconds beyond control)).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1993-06; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kuo G, Choo QL, Alter HJ, Gitnick GL, Redeker AG, Purcell RH, Miyamura T, Dienstag JL, Alter MJ, Stevens CE, et al. An assay for circulating antibodies to a major etiologic virus of human non-A, non-B hepatitis. Science. 1989 Apr 21;244(4902):362-4. doi: 10.1126/science.2496467.
- [Background] Alter MJ, Margolis HS, Krawczynski K, Judson FN, Mares A, Alexander WJ, Hu PY, Miller JK, Gerber MA, Sampliner RE, et al. The natural history of community-acquired hepatitis C in the United States. The Sentinel Counties Chronic non-A, non-B Hepatitis Study Team. N Engl J Med. 1992 Dec 31;327(27):1899-905. doi: 10.1056/NEJM199212313272702. PMID 1280771